CLINICAL TRIAL: NCT00006117
Title: Phase II Study of Gemcitabine Plus Oxaliplatin in Patients With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Gemcitabine and Oxaliplatin in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068130; FRE-GERCOR-GEMOX-D99-2; EU-20027
Record Dates: First submitted 2000-08-03; First posted 2004-06-22 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; stage IV pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine and oxaliplatin in treating patients who have locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective tumor response rate in patients with locally advanced or metastatic pancreatic carcinoma when treated with gemcitabine and oxaliplatin. II. Determine the tolerablility and clinical benefit of this regimen in these patients. III. Evaluate the progression free survival and the overall survival of these patients when treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive gemcitabine IV on day 1 over 1.5 hours and oxaliplatin IV over 2 hours on day 2. Treatment continues every 2 weeks in the absence of disease progression or unacceptable toxicity. Patients with locally advanced disease receive 6-8 courses and then may undergo surgery, radiotherapy, and/or additional chemotherapy.

PROJECTED ACCRUAL: A total of 66 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed metastatic or locally advanced unresectable adenocarcinoma of the pancreas Measurable disease At least 2 cm in diameter No known brain metastases

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance status: ECOG 0-2 OR Karnofsky 60-100% Life expectancy: Greater than 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 5 times ULN Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: Adequate cardiac function Pulmonary: Adequate respiratory function Other: Not pregnant or nursing Fertile patients must use effective contraception No sensitive neuropathy No other active malignancy No uncontrolled hypercalcemia No significant medical or psychiatric condition that would preclude study No psychological, familial, sociological, or geographical condition that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy Chemotherapy: No prior chemotherapy Endocrine therapy: No concurrent corticosteroid use except as antiemetic Radiotherapy: No prior radiotherapy Surgery: Not specified Other: No other concurrent investigational drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Louvet, MD, PhD, Study Chair — Hopital Saint Antoine
Locations (10):
- Institut Jules Bordet, Brussels, Belgium
- France (9):
  - Centre Paul Papin, Angers
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Hopital Beaujon, Clichy
  - Hopital Drevon, Dijon
  - Clinique Saint Jean, Lyon
  - American Hospital of Paris, Neuilly-sur-Seine
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Polyclinique De Courlancy, Reims

REFERENCES:
- [Background] Huguet F, Andre T, Hammel P, Artru P, Balosso J, Selle F, Deniaud-Alexandre E, Ruszniewski P, Touboul E, Labianca R, de Gramont A, Louvet C. Impact of chemoradiotherapy after disease control with chemotherapy in locally advanced pancreatic adenocarcinoma in GERCOR phase II and III studies. J Clin Oncol. 2007 Jan 20;25(3):326-31. doi: 10.1200/JCO.2006.07.5663. PMID 17235048
- [Result] Afchain P, Chibaudel B, Lledo G, Selle F, Bengrine-Lefevre L, Nguyen S, Paitel JF, Mineur L, Artru P, Andre T, Louvet C. First-line simplified GEMOX (S-GemOx) versus classical GEMOX in metastatic pancreatic cancer (MPA): results of a GERCOR randomized phase II study. Bull Cancer. 2009 May;96(5):E18-22. doi: 10.1684/bdc.2009.0871. Epub 2009 May 12. PMID 19435690
- [Result] Louvet C, Andre T, Lledo G, Hammel P, Bleiberg H, Bouleuc C, Gamelin E, Flesch M, Cvitkovic E, de Gramont A. Gemcitabine combined with oxaliplatin in advanced pancreatic adenocarcinoma: final results of a GERCOR multicenter phase II study. J Clin Oncol. 2002 Mar 15;20(6):1512-8. doi: 10.1200/JCO.2002.20.6.1512. PMID 11896099